# Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic Lesions on 18F-FDG-PET/CT in Head and Neck Squamous Cell Carcinoma

NCT05747625

Document Date: August 1, 2025

IRB Approval Date: August 7, 2025

Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma 08/01/2025

PI: Michael Topf, MD, MSCI

Version Date:

| Name of participant: | Age: |
|----------------------|------|

The following is given to you to tell you about this research study. Please read this form with care and ask any questions you may have about this study. Your questions will be answered. Also, you will be given a copy of this consent form.

#### **Key Information:**

The first section of this document contains some key points that the research team thought you would find important. The study is described in more detail after this section. If you do not understand something, please ask someone.

### **Key information about this study:**

#### **General Information**

You are invited to participate in a research study to determine the diagnostic utility of <sup>89</sup>Zr-panitumumab to identify metastatic and/or primary lesion(s) in subjects with head and neck squamous cell carcinoma (HNSCC). You were selected because it was found that you have indeterminate lesions on routine Positron Emission Tomography (PET) scans of lesion metabolism (18F-FDG-PET) and computed tomography (CT) scans of lesion structure and are scheduled to undergo further evaluation of the lesions per standard of care.

This research study is looking for 60 participants with HNSCC. Vanderbilt University is the only site to participate in the study and expects to enroll all 60 research study participants.

You should not feel obligated to agree to participate. Your questions should be answered clearly and to your satisfaction. If you decide not to participate, please tell the Protocol Director.

### **Purpose**

We hope to determine if PET imaging using a new radiotracer named (89Zr)-panitumumab, which can bind to tumors and enable these tumors to be visualized, can help us to better identify tumors compared to the information obtained from standard measures of metabolism and tissue structure obtainable from more common imaging methods, such as PET, magnetic resonance imaging (MRI), and computed tomography (CT). Before 1-5 days of the scan, you will also receive the drug, panitumumab which is an FDA approved chemotherapy agent for treating other types of






Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma

Version Date: 08/01/2025

PI: Michael Topf, MD, MSCI

cancer such as colon cancer. The total dose of panitumumab that you will receive will be lower than the usual total dose that is given to patients receiving it as a treatment for cancer.

### **Voluntary Participation**

Your participation in this study is entirely voluntary. Your decision not to participate will not have any negative effect on you or your medical care. You can decide to participate now but withdraw your consent later and stop being in the study without any loss of benefits or medical care to which you are entitled. If we learn something new that may affect the risks or benefits of this study, you will be told so that you can decide whether or not you still want to be in this study. Your medical record will contain a note saying you are in a research study and may contain some research information about you. Anyone you authorize to receive your medical record will also get this information.

### **Duration & Visits**

Your participation in this research study is expected to take approximately 45 days, with up to 30 days for screening to see if you are eligible to participate (screening period can be shorter than 30 days) and approximately 15 days on study. You will only have 2-3 research specific visits, in addition to your normal imaging and follow-up clinic visits and examinations.

There is a 36-month (± 6 months) data collection point after your active participation for information about the status of your indeterminate lesion(s) only through review of your electronic medical records. There will be no visits required.

#### **Overview of Procedures**

If you agree to enroll, you will receive a one-time injection of both panitumumab and <sup>89</sup>Zr panitumumab 1 - 5 days before receiving a PET/CT scan. You will be evaluated for any reactions to the drug immediately after the injection and up to 15 days after the scan.

### **Risks**

The most likely risks are infusion reactions, rash, dry or itchy skin, fatigue, decreased magnesium and/or other minerals in your blood, and radiation exposure.

#### **Benefits**

You may or may not have a direct benefit from being in the study. But the study doctors hope to be able to use the information on the safety of the radiotracer to help treat future cancer patients.






Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

#### **Alternatives**

This study is in the setting of tumor excision of biopsy confirmed diagnosis of HNSCC, and the experimental component is infusion of 89Zrpanitumumab, which may help visualize the tumor and identify tumor loaded lymph nodes. The alternative to participating in this study is to not participate in the trial.

#### **Detailed Information:**

The rest of this document includes detailed information about this study (in addition to the information listed above).

You are being asked to take part in this research study because it was found that you have indeterminate lesions on a routine <sup>18</sup>F-FDG-PET/CT preoperative imaging and are scheduled to undergo further evaluation of the lesions per standard of care.

Indeterminate lesions are broadly defined as lesions that cannot be confidently characterized as either positive or negative and require further clarification through discussion at a multidisciplinary meeting, planned further investigation, or intervention.

You do not have to be in this research study. You may choose not to be in this study and get other treatments without changing your healthcare, services, or other rights. You can stop being in this study at any time. If we learn something new that may affect the risks or benefits of this study, you will be told so that you can decide whether or not you still want to be in this study. Your medical record will contain a note saying you are in a research study and may contain some research information about you. Anyone you authorize to receive your medical record will also get this information.

### Side effects and risks that you can expect if you take part in this study:

There are risks, discomforts, and inconveniences associated with any research study. These deserve careful thought. You should talk with the Protocol Director if you have any questions.

### Potential Risks of Panitumumab (VECTIBIX ®)

<sup>89</sup>Zr panitumumab contains the panitumumab antibody. Panitumumab is approved by the US FDA for treatment of certain types of advanced colorectal cancer at a dosage of 6 mg/kg given every 14 days. Many of the reported adverse events are associated with repeat administration of panitumumab, rather than the single dose that you will receive as part of this study. The total dose of panitumumab that you will receive will be lower than the usual total dose that is given to patients receiving it as treatment for cancer.


**Institutional Review Board** 

**VANDERBILT** 

Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

The most common side effects patients have experienced when receiving panitumumab primarily include skin reactions (including acne like rash, dry or itchy skin, cracking of skin around your nail beds, skin infections, and dry eyes), fatigue, nausea, and diarrhea. Monitor skin reactions carefully to prevent serious or life-threatening complications. Exposure to sunlight may make skin reactions worse; limit exposure by using sunscreen and protective clothing.

Infusion reactions, including fever, chills, difficulty or labored breathing, and low blood pressure, occurred in 4% of patients taking panitumumab. These reactions are most likely during or immediately following panitumumab infusion. Severe infusion reactions occurred in 1% of patients. Based on your study doctor's routine practice, he or she may decide to give other drugs, such as an antihistamine called diphenhydramine (Benadryl) or steroids, if it's felt necessary to treat a reaction. Tell your doctor or nurse immediately if you experience any of the ymptoms of an infusion reaction.

Patients receiving repeated doses of panitumumab occasionally had progressively decreased magnesium and/or other minerals in the blood. Your blood chemistry levels will be monitored closely during this study, and electrolyte replacement will be given if necessary.

There have been rare reports of patients experiencing fatal and non-fatal lung disease after treatment with panitumumab. You should notify your study doctor if you have ever had lung disease. *Tell your doctor or nurse immediately if you experience* sudden or worsening breathing troubles.

# Potential Risks of 89Zr panitumumab

The expected risks of <sup>89</sup>Zr panitumumab are expected to be the same as the known risks of panitumumab (see above section) and the additional risks of the <sup>89</sup>Zr chelator, deferoxamine (DFO).

We use DFO to help us link together panitumumab and Zirconium. As a result, DFO is found in the solution containing the study agent, 89Zr panitumumab.

Deferoxamine is approved by the US FDA and throughout much of the world for the treatment of acute iron intoxication and of chronic iron overload due to transfusion dependent anemias. Deferoxamine is a metal chelator, meaning it binds to a metal atom (in this case, Zirconium-89). The most likely possible side effects of deferoxamine include localized reactions at the site of IV placement, including irritation, pain; burning; swelling; induration (hardening of the skin); itching; redness; rash or scabbing of the skin.






Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

In addition to injection site reactions, deferoxamine can also cause an allergic or hypersensitivity reaction in your body. Symptoms of a systemic (whole body) allergic reaction include rash, hives, anaphylactic reaction, swelling or tightness of the face or throat, nausea, vomiting, diarrhea, dizziness or fainting, fast heartbeat, and/or low blood pressure. *Tell your doctor or nurse immediately if you experience any of the symptoms of an allergic reaction.* 

We do not believe that the radiotracer will increase your chances of experiencing known side effects from treatment with panitumumab; however, we do not know this for sure. The most common dose independent side effects associated with panitumumab are infusion reaction or allergic reactions, described in the panitumumab risk section above. <sup>89</sup>Zr panitumumab is radioactive, so you will be exposed to radiation from the radiotracer. The radiation risks are discussed in a separate section below.

### **Radiation Risks:**

You are agreeing to participate in a research project that involves the use of imaging procedures that expose you to radiation. This section will discuss the risks associated with the imaging procedures that are for research only. Your doctors may order additional imaging procedures as part of your normal patient care that also expose you to radiation. Those normal imaging procedures are not included in the risk discussion below. Please discuss those procedures and radiation risks with your doctors. As part of this research study, you may be asked to have an additional imaging procedure that exposes you to radiation. This procedure is known as a PET-CT scan (Positron Emission Tomography-Computed Tomography). It exposes you to external radiation from the CT portion as well as internal exposure from injection of a radioactive substance. The amount of radiation that you could receive from this total procedure is approximately 49-98% of the amount allowed annually for persons who are exposed to radiation as part of their work. Additionally, to protect your bladder from the effects of the injected radioactive substance, you should drink plenty of fluids and empty your bladder every two hours for at least the first six hours after you have the PET/CT scan.

### **Potential Reproductive Risks**

### Women of Childbearing Potential

Based on data from animal studies, panitumumab may cause fetal harm (organ damage, death) when administered to pregnant women. If you are a woman who is able to become pregnant, it is expected that you will use an effective method of birth control to prevent exposing a fetus to a potentially dangerous agent with unknown risk. If you are pregnant or currently breast feeding, you may not participate in this study. You understand that if you are pregnant, if you become pregnant, or if you are breast feeding during this study, you or your child may be exposed to an unknown risk.




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

### **Potential Study Procedure Risks**

Blood Draw/IV: Inserting a needle into your arm for drawing blood, or an IV catheter for infusion, can cause slight discomfort or bruising at the puncture site. Lightheadedness or fainting may occur. Rarely, an infection at the puncture site may occur.

### Risks that are not known:

Because this study is investigational, meaning non-FDA approved, there may be risks that we do not know about at this time.

### Benefits that might result from this study:

You may not benefit directly from taking part in this study. However, information obtained from your participation in this study may benefit other people with cancer in the future and help determine if <sup>89</sup>Zr panitumumab can be used as an alternative for the current standard treatments for the preoperative identification of lesion(s) of HNSCC.

We cannot and do not guarantee or promise that you will receive any benefits from this study.

#### Procedures to be followed:

If you choose to participate in this study, the Protocol Director and their research team will perform the procedures listed below in addition to your normal pre-operative, surgery and follow up clinic visits and examinations. Please refer to Table 1.




Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic and/or Primary Lesions on 18F-FDG-PET/CT in Head and Neck Squamous Cell Study Title:

Carcinoma

08/01/2025 Version Date:

PI: Michael Topf, MD, MSCI

Table 1: Study Calendar for all visit specific procedures.

| Table 1: Study Calendar for all visit specific procedures. Table 1: Study Calendar | | | | | |
|---|---|---|---|---|---|
| STUDY VISIT PROCEDURES | SCREENING/ PRETREATMENT (WITHIN 30 DAYS OF START OF TREATMENT) | Day<br>0 | Day 1<br>TO 5 | DAY 15<br>(± 7 DAYS) | STANDARD<br>OF CARE<br>FOLLOW-<br>UP |
| INFORMED CONSENT | X | | | | |
| MEDICAL HISTORY | X | | | | |
| VITAL SIGNS | Х | Χ | | | |
| PHYSICAL EXAMINATION | Х | | | | |
| CLINICAL ASSESSMENT | | | | Х | |
| PERFORMANCE STATUS (ECOG) | Х | | | | |
| ECG | Х | Χ | | Х | |
| CLINICAL CHEMISTRIES | Х | | | | |
| HEMATOLOGY | Х | | | | |
| SERUM PREGNANCY | Х | | | | |
| URINE PREGNANCY | | Х | | | |
| COLLECTION OF PREVIOUS <sup>18</sup> F-<br>FDG PET/CT IMAGING DATA FROM<br>MEDICAL RECORD | Х | | | | |
| Unlabeled Panitumumab<br>Infusion | | X | | | |
| BOLUS INJECTION OF 89ZR<br>PANITUMUMAB | | Х | | | |
| 89ZR TUMOR IMAGING | | | Х | | |
| ADVERSE EVENTS | Χ | X | Х | Х | |
| CONCOMITANT MEDICATIONS | Х | Χ | X | Х | |
| STANDARD OF CARE EVALUATION OF LESIONS | | | | х | х |
| CHART REVIEW OF SUBJECTS | | | | | Χ |




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

### **Screening Period**

If you choose to participate in the study and sign this consent form, you will have to undergo the following exams and tests to determine if you are eligible to take part in this study. If you have already had some of these exams (physical exam, performance status, and vital signs) and tests (blood work for clinical Chemistries and Hematology) recently, they may not need to be repeated. The screening period will not last more than 30 days.

The following procedures will occur during **Screening**:

- Review your medical history and current medications.
- Physical exam, including height, weight, and vital signs (blood pressure, heart rate, respiratory rate, and temperature).
- Performance status a measure of how you are feeling.
- Electrocardiogram (ECG) a test to measure and record the electrical activity of your heart.
   Sticky pads will be placed at different points on your body, and you will be asked to lie still while the machine records your heart activity.
- Blood draw for lab safety tests (approximately 2 teaspoons).
- Pregnancy test if you are a woman who could have children (approximately ½ teaspoon of blood); if you are pregnant or breast feeding you cannot participate in this study because of the potential unknown risk to your unborn fetus or baby. And please ensure use of effective contraception during screening and to be continued for 2 months following administration of panitumumab and 89Zr-panitumumab doses.
- Assessment of side effects (adverse events) related to study
- Obtain a copy of results from an <sup>18</sup>F FDG PET/CT scan and/or other available images that are part of your standard of care pre-operative tests.

### Day 0

If you meet all the requirements to participate, you will come to clinic on Day 0 to receive the investigational imaging agent. The following procedures will occur:

### Prior to ANY drug administration:

- A pregnancy test for women of childbearing potential will be required, and please ensure use of effective contraception during screening and to be continued for 2 months following administration of panitumumab and 89Zr-panitumumab doses.
- Vital signs (blood pressure, heart rate, pulse oximetry, respiratory rate)
- o FCG
- Assessment for concomitant medications




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma 08/01/2025

Pl: Michael Topf, MD, MSCI

Version Date:

- Administration of unlabeled panitumumab: The agent will be given as a single dose over 15 minutes (± 5 minutes) through an IV tube into a vein in your arm followed by:
  - Observation for 30 minutes (± 10 minutes)
    - Safety monitoring for 30 minutes after the end of the study agent administration to watch for side effects. Your study doctor may prescribe other medications to treat or prevent side effects. At any time during this treatment, it is important for you to let your doctor or nurse know if you experience anything that does not feel normal.
  - o Assessment for side effects (adverse events) at the end of observation period
  - Vital signs (blood pressure, heart rate, pulse oximetry, respiratory rate)
  - o ECG
- Prior to injection of 89Zr-panitumumab:
  - Vital signs (blood pressure, heart rate, pulse oximetry, respiratory rate)
- Administration of <sup>89</sup>Zr-panitumumab: The study agent will be given as a single dose given all at once through the IV tube into a vein in your arm, followed by:
  - Vital signs (blood pressure, heart rate, pulse oximetry) approximately 15 minutes (±10 minutes) after injection of 89 Zrpanitumumab
  - Observation for 30 minutes (± 10 minutes)
    - Safety monitoring for 30 minutes after the end of the study agent administration to watch for side effects. Your study doctor may prescribe other medications to treat or prevent side effects. At any time during this treatment, it is important for you to let your doctor or nurse know if you experience anything that does not feel normal.
  - Assessment for side effects (adverse events) at the end of observation period
  - Assessment for medications you are taking at the time

#### DAY 1 TO DAY 5:

On Day 1 to Day 5, depending on schedule availability, you will be asked to come to clinic to have your <sup>89</sup>Zrpanitumumab PET/CT imaging. This visit will include:

- PET/CT imaging: During image collection, study doctors will collect both head through abdomen PET images, which detect the small amount of radiolabeled <sup>89</sup>Zrpanitumumab imaging agent, and CT images, which uses X-rays, to look at your tissues and organs. You will be asked to lie on a long narrow couch for up to 90 minutes while the machine gathers
- An assessment for any side effects and review current medications.


**Institutional Review Board** 

**VANDERBILT** 

Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

### Day 15:

On Day 15, a clinical assessment will be performed in-person or via telehealth to include collection of any side effects that are attributable to the study and/or a review of current medications. You may also receive an ECG if it is medically indicated.

### **Continuation of standard of care:**

You will resume standard of care treatment as previously determined by your treatment team. The study will not impact the standard of care treatment you receive.

### Follow-up:

You will be followed for  $36 \pm 6$  months, with possibility for extension, via external chart review to compare  $^{89}$ Zr-PET/CT results to standard of care follow-up. You will not be asked to make any in-person or telehealth visits during this time, nor will you have any contact with the study during this time.

### **Specimen Storage for Future Research**

Research using human specimens is an important way to try to understand human disease. You have been given this information because the investigators will save your specimens including oral swabs, blood and tissue for future research if they are available from your standard of care and as standard of procedure for the Head and Neck Repository. There are several things we would like you to be informed about.

Your specimens and any data collected as part of this study will be stored in the Head and Neck Biorepository (IRB# 030062) at Vanderbilt University Medical Center (VUMC). Samples will be labeled with a study ID code number that does not personally identify you.

The key linking the study ID code with your personal information will not be shared with researchers. Your samples may be sent outside of VUMC for research and analysis. Identifiers will be removed from identifiable private information and/or identifiable specimens, and, after such removal, the information and/or specimens could be used for future research studies or distributed to investigators within or outside VUMC for future research studies without additional informed consent from you.

### Monetary compensation for your time spent taking part in this study or expenses:

You may receive up to a total \$200 if you complete this study. You will be paid for the visits you completed according to the following schedule:

•\$100 for the Infusion Day Visit •\$100 for the Imaging Visit


**Institutional Review Board** 

**VANDERBILT** 

Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

If you do not complete the study, for any reason, you will be paid for each study visit you do complete. We will complete a check request for you via Vanderbilt's Finance Department at the end of your participation. The check may take 4-6 weeks to process. We may ask you for your Social Security number and address on a form before you are compensated for taking part in the study.

In addition to monetary compensation, you will receive travel reimbursement up to \$600 total with appropriate receipts and/ or documentation to study team.

If you have any questions regarding your compensation for participation, please contact the study staff.

### Costs to you if you take part in this study:

If you agree to take part in this research study, you and/or your insurance will not have to pay for the tests and treatments that are being done only for research. However, you are still responsible for paying for the usual care you would normally receive for the treatment of your illness. This includes treatments and tests you would need even if you were not in this study. These costs will be billed to you and/or your insurance.

You have the right to ask what it may cost you to take part in this study. If you would like assistance, financial counseling is available through the Vanderbilt Financial Assistance Program. The study staff can help you contact this program. You have the right to contact your insurance company to discuss the costs of your routine care (non-research) further before choosing to be in the study. You may choose not to be in this study if your insurance does not pay for your routine care (non-research) costs and your doctor will discuss other treatment plans with you.

### Payment in case you are injured because of this research study:

If it is determined by Vanderbilt and the Investigator, Dr. Michael Topf, that an injury occurred as a direct result of the tests or treatments that are done for research, then you and/or your insurance will not have to pay for the cost of immediate medical care provided at Vanderbilt to treat the injury.

There are no plans for Vanderbilt or Dr. Michael Topf to pay for any injury caused by the usual care you would normally receive for treating your illness or the costs of any additional care. There are no plans for Vanderbilt or Dr. Michael Topf to give you money for the injury.




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma 08/01/2025

Pl: Michael Topf, MD, MSCI

Version Date:

### Who to call for any questions or in case you are injured:

If you should have any questions about this research study or if you feel you have been hurt by being a part of this study, please feel free to contact the study doctor. You may contact Dr. **Michael Topf** at **(585) 278-4883**. Your study coordinator will also provide you with contact information. If you cannot reach the research staff, please page the study doctor (Dr. Michael Topf) by calling (615) 322-5000 and ask the operator to page him.

For additional information about giving consent or your rights as a person in this study, to discuss problems, concerns, and questions, or to offer input, please feel free to call the VUMC Institutional Review Board Office at (615) 322-2918 or toll free at (866) 224-8273.

### Reasons why the study doctor may take you out of this study:

The Protocol Director may also withdraw you from the study and administration of the study agent may be stopped without your consent for one or more of the following reasons:

- Failure to follow the instructions of the Protocol Director and study staff.
- The Protocol Director decides that continuing your participation could be harmful to you.
- Pregnancy
- You need treatment not allowed in the study.
- The study is cancelled.
- Other administrative reasons.
- Unanticipated circumstances.

### What will happen if you decide to stop being in this study?

If you first agree to participate and then you change your mind, you are free to withdraw your consent and discontinue your participation at any time. Your decision will not affect your ability to receive medical care for your disease and you will not lose any benefits to which you would otherwise be entitled.

If you withdraw from the study, or administration of the study agent is stopped for any reason, you will be asked to return to the clinic approximately one month from Day 0 for a safety follow up appointment (will be coordinated where possible with a routine visit).

### **Clinical Trials Registry:**

A description of this clinical trial will be available on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

### **Confidentiality:**

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed except as authorized by you or as required by law. However, there is always some risk that even de-identified information might be re-identified.

Patient information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

The purpose of this research study is to obtain information on the safety and effectiveness of <sup>89</sup>Zr-panitumumab. The results will be provided to the sponsor, the Food and Drug Administration and other federal and regulatory agencies as required.

This study will utilize Research Electronic Data Capture (REDCap), a software toolset and workflow methodology for electronic collection and management of clinical and research data, to collect and store data. REDCap was developed specifically around HIPAA Security guidelines. The system includes password protection and internal quality checks.

Your excess tissue samples for future research if they are available from your standard of care will be stored in a Tissue Repository at Vanderbilt University Medical Center (VUMC). Samples will be labeled with a study ID code number that does not personally identify you. Identifiers will be removed from identifiable private information and/or identifiable specimens, and, after such removal, the information and/or specimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you.

Only the investigator(s) and authorized study team members have the access to your data and specimens. And these materials will be made available for monitoring and/or auditing by Medical Monitor, other monitoring body and/or regulatory agencies.

This study may have some support from the National Institutes of Health (NIH). If so, your study information is protected by a Certificate of Confidentiality. This Certificate allows us, in some cases, to refuse to give out your information even if requested using legal means.

It does not protect information that we have to report by law, such as child abuse or some infectious diseases. The Certificate does not prevent us from disclosing your information if we learn of possible harm to yourself or others, or if you need medical help.




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

Disclosures that you consent to in this document are not protected. This includes putting research data in the medical record or sharing research data for this study or future research. Disclosures that you make yourself are also not protected.

### Privacy:

Any radiological imaging and information about you may be made available to others to use for research. To protect your privacy, we will not release your name. You will not receive any benefit as a result of the tests done on you. These tests may help us, or other researchers learn more about the causes, risks, treatments, or how to prevent this and other health problems.

### **Study Results:**

The research results will be shared with you when the study is closed out by request. The shared study results may include peer-reviewed scientific publications, news releases, and clinical trials reports at ClinicalTrials.gov.

#### Authorization to Use/Disclose Protected Health Information

## What information is being collected, used, or shared?

To do this research, we will need to collect, use, and share your private health information. By signing this document, you agree that your health care providers (including both Vanderbilt University Medical Center and others) may release your private health information to us, and that we may use any and all of your information that the study team believes it needs to conduct the study. Your private information may include things learned from the procedures described in this consent form, as well as information from your medical record (which may include information such as HIV status, drug, alcohol or STD treatment, genetic test results, or mental health treatment).

### Who will see, use or share the information?

The people who may request, receive or use your private health information include the researchers and their staff. Additionally, we may share your information with other people at Vanderbilt, for example if needed for your clinical care or study oversight. By signing this form, you give permission to the research team to share your information with others outside of Vanderbilt University Medical Center. This may include the sponsor of the study and its agents or contractors, outside providers, study safety monitors, government agencies, other sites in the study, data managers and other agents and contractors used by the study team. We try to make sure that everyone who sees your information keeps it confidential, but we cannot guarantee that your information will not be shared with others. If your information is disclosed by your health






Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma


PI: Michael Topf, MD, MSCI

care providers or the research team to others, federal and state confidentiality laws may no longer protect it.

### Do you have to sign this Authorization?

You do not have to sign this Authorization, but if you do not, you may not join the study.

## How long will your information be used or shared?

Your Authorization for the collection, use, and sharing of your information does not expire. Additionally, you agree that your information may be used for similar or related future research studies.

### What if you change your mind?

You may change your mind and cancel this Authorization at any time. If you cancel, you must contact the Principal Investigator in writing to let them know by using the contact information provided in this consent form. Your cancellation will not affect information already collected in the study, or information that has already been shared with others before you cancelled your authorization.

### Michael Topf, MD, MSCI

Vanderbilt University Medical Center 7320 Medical Center East, South Tower 1215 21st Avenue South, Nashville, TN 37232

If you decide not to take part in this research study, it will not affect your treatment, payment or enrollment in any health plans or affect your ability to get benefits. You will get a copy of this form after it is signed.




Study Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic

and/or Primary Lesions on <sup>18</sup>F-FDG-PET/CT in Head and Neck Squamous Cell

Carcinoma 08/01/2025

Pl: Michael Toof M

PI: Michael Topf, MD, MSCI

## STATEMENT BY PERSON AGREEING TO BE IN THIS STUDY

I have read this consent form and the research study has been explained to me verbally. All my questions have been answered, and I freely and voluntarily choose to take part in this study.

| Date | Signature of patient/volunteer |
|----------------------|--------------------------------|
| Consent obtained by: | |
| Date | Signature |
| | Printed Name and Title |


